CLINICAL TRIAL: NCT07233772
Title: The Effect of a Motivational Interviewing-Based Constipation Training Program Given to Mothers on Maternal Anxiety Levels and Children's Constipation Symptoms: A Randomized Controlled Trial
Brief Title: Effect of Motivational Interviewing Training on Mothers' Anxiety and Children's Constipation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Kübra Koçyiğit Gültepe, PhD Candidate, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: necmettineu-koçyiğitgültepe-01
Record Dates: First submitted 2025-09-29; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Function Constipation; Anxiety
Keywords: children; functional constipation symptoms; education program; maternal anxiety; motivational interviewing
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This study uses a parallel assignment model. Participants will be randomly assigned to either the intervention group, which will receive a motivational interview-based constipation education program, or the control group, which will receive no intervention. Randomization will be performed using a block randomization method to ensure balanced allocation between groups. Outcomes will be compared at the end of the intervention period
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): First, the researcher will introduce herself and explain the purpose of the study to the participants. Pre-tests will be administered to individuals who meet the inclusion criteria and agree to participate in the study. At the pre-test stage, the Mother and Child Descriptive Information, Defecation Frequency, Bristol Stool Form Scale, and Trait Anxiety Inventory will be administered. During follow-up assessments, Defecation Frequency and the Bristol Stool Form Scale will be used. At the final follow-up, Defecation Frequency, the Bristol Stool Form Scale, and the Trait Anxiety Inventory will be administered. A motivational interviewing-based intervention program will be implemented for the intervention group, and the follow-up period will last for one month.
  Interventions: Other: Motivational Interview-Based Constipation Education Program
- Control Group (No Intervention): In the study, no intervention will be applied to the mothers in the control group. As stated prior to the study, after the post-test data are collected, training will be planned for the participants in the control group and the training materials will be provided. At the pre-test stage, the Mother and Child Descriptive Information Form, Defecation Frequency, Bristol Stool Form Scale, and Trait Anxiety Inventory will be administered. During follow-ups, Defecation Frequency and the Bristol Stool Form Scale will be used. At the post-test stage, Defecation Frequency, the Bristol Stool Form Scale, and the Trait Anxiety Inventory will be administered. The follow-up period will last for one month.

INTERVENTIONS:
Other: Motivational Interview-Based Constipation Education Program — Structured educational sessions delivered to mothers using motivational interviewing techniques, aiming to reduce maternal anxiety and improve children's constipation symptoms
  Arms: Intervention Group

SUMMARY:
Study Description (Brief Summary) Functional constipation (FC) is one of the most common gastrointestinal disorders in children. It is a widespread bowel condition characterized by persistent difficulty, incomplete, or infrequent defecation without an organic, endocrine, or metabolic cause. The prevalence of functional constipation in childhood ranges between 5% and 30%. The preschool period is considered a risk factor for functional constipation, as children experience new beginnings and spend extended time away from home due to school. During this period, mothers may experience increased anxiety. The aim of this study is to reduce maternal anxiety and improve children's constipation symptoms through a constipation training program based on motivational interviewing delivered to mothers.

DETAILED DESCRIPTION:
Constipation is a common problem in children and can cause discomfort and anxiety for both the child and the family. This study aims to help mothers manage their children's constipation symptoms through a training program based on motivational interviewing. The program focuses on improving mothers' knowledge, motivation, and confidence in supporting their children's healthy bowel habits. The study also examines whether this approach reduces mothers' anxiety levels. The results are expected to contribute to better management of constipation in children and improved family well-being.

ELIGIBILITY:
Inclusion Criteria:

Mother of a 4-6 year old child attending preschool/kindergarten with functional constipation diagnosed per Rome IV criteria

Exclusion Criteria:

Mothers of children with congenital anomalies or chronic gastrointestinal disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2025-11-24 (Estimated); Study Completion 2025-12-22 (Estimated)

PRIMARY OUTCOMES:
Defecation Frequency | From baseline to the end of the fourth week, with assessments conducted at the end of the first, second, third, and fourth weeks.
  The number of defecations per week will be recorded to assess changes in bowel movement frequency during the study. According to the Rome IV criteria, the weekly defecation frequency must be more than two times per week in order not to be classified as functional constipation.
Bristol Stool Form Scale (BSFS) | From baseline to the end of the fourth week, with assessments conducted at the end of the first, second, third, and fourth weeks.
  Stool consistency will be assessed using the Bristol Stool Form Scale to evaluate changes over the intervention period. Seven stool types are classified. Types 1 and 2 (scores 1 and 2) indicate hard stools, which are associated with constipation; Types 3, 4, and 5 (scores 3, 4, and 5) represent normal stool forms; and Types 6 and 7 (scores 6 and 7) indicate loose or watery stools, typically observed in diarrhea.

SECONDARY OUTCOMES:
Trait Anxiety Inventory (STAI-T) | From baseline to the end of the fourth week, with assessments conducted at the end of the first and fourth weeks.
  Maternal trait anxiety will be assessed using the Trait Anxiety Inventory Form. The change in scores from baseline to post-intervention will be analyzed. The total score obtained from the scale ranges from 20 to 80. Higher scores indicate higher levels of anxiety, whereas lower scores indicate lower levels of anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Preschools Affiliated with the Ministry of National Education, Karaman, Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data (IPD) in order to ensure the protection of participants' personal information and confidentiality.